CLINICAL TRIAL: NCT00057226
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Flexible-Dose Study Evaluating Efficacy, Safety, and Tolerability of Once-Daily Oral GW353162 (40-60mg) Versus Placebo in Subjects With Major Depressive Disorder Over an Eight-Week Treatment Period.
Brief Title: An 8 Week Study Of Adults Diagnosed With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHB20003
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Depressive Disorder, Major
Keywords: GW353162,; Major depressive disorder,; flexible
MeSH Terms: conditions — Depressive Disorder, Major | interventions — radafaxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Radafaxine

SUMMARY:
A Placebo Controlled Study Evaluating Efficacy, Safety and Tolerability of Medication in Patients with Major Depressive Disorder (MDD)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD)
* Duration of current depressive episode 12 weeks - 24 months
* Patients can read and write at a level sufficient to provide a signed consent
* If female, patients must be practicing an acceptable method of birth control

Exclusion Criteria:

* Patients have other psychiatric disorders that would affect patient's response to treatment
* Patients have not responded to two or more adequate courses of antidepressant therapy
* Patients cannot be currently abusing illicit drugs or alcohol
* Patients are not currently receiving psychotherapy
* Patients have received electroconvulsive therapy within 6 months prior to screening
* Patients are pregnant or lactating

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2003-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) score after 8 weeks of treatment | 8 Weeks

SECONDARY OUTCOMES:
Change in the MADRS score at other timepoints; change in the Global Impression; percentage of remitters and responders based on the MADRS; change in anxiety, disability, motivation, energy, fatigue and pain; incidence of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Libertyville, Illinois
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Bellevue, Washington